CLINICAL TRIAL: NCT01450852
Title: Strength Training Induced Alterations in Markers of Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Laura Stewart, Assistant Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LSU-IRB # 3005
Record Dates: First submitted 2011-10-03; First posted 2011-10-12 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Inflammation
Keywords: Melanocortin Receptor; Monocyte; Resistance Training; Inflammation; Markers of Inflammation
MeSH Terms: conditions — Inflammation | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strength Training (Experimental): The strength training group completed 12 weeks of progressive, periodized resistance training 3d/wk.
  Interventions: Behavioral: Strength Training
- Active Control Group (No Intervention): The active control group was instructed to maintain normal activity and eating habits. They participated in all pre and post intervention measures.

INTERVENTIONS:
Behavioral: Strength Training — Each Member of this group completed 12 weeks of progressive, periodized resistance training for 3d/wk.
  Arms: Strength Training

SUMMARY:
Exercise has been used to help prevent or slow the progression of inflammation-related disease; however, the mechanism by which this activity may lower concentrations of inflammatory markers remains unclear. The melanocortin receptors 1,3 and 5 (MC1R, MC3R and MC5R) have been shown to function in an anti-inflammatory manner and have the potential to mediate the positive immune adaptations associated with regular physical activity.

Preliminary data suggest that MC3R gene expression increases in whole blood after chronic exercise training. The primary aim of the current study is to explore whether this change in gene expression translates into alterations in MC1R, MC3R, or MC5R monocyte surface expression. The secondary aim is to examine the relationship between surface expression of these receptors and circulating inflammatory profiles.

The investigators will recruit 42 untrained, healthy males and females aged 18-35 yrs. Half of the group will be placed on an exercise program for 15 weeks. The other half will serve as untrained control subjects. In addition to basic anthropometric measures, the investigators will measure concentrations of inflammatory and anti-inflammatory cytokines (ELISA) and cell surface expression of MC1R, MC3R, and MC5R on monocytes (flow cytometry).

DETAILED DESCRIPTION:
Abstract:

Chronic exercise reduces inflammation, but the mechanisms involved are unclear. Recent studies have shown that stimulation of melanocortin 1 and 3 receptors (MC1R and MC3R) on immune cells increases anti-inflammatory cytokine production. PURPOSE: To examine the influence of 12 weeks of resistance training (RT) on body composition, monocyte cell-surface expression of MC1R and MC3R and circulating markers of inflammation. METHODS: Healthy, active males and females (age 20-27 yr) were recruited into a RT group (RE; n = 23) and an active control group (AC; n = 19). RE completed 12 weeks of progressive, periodized RT 3d/wk while AC maintained normal activity habits. Measures of body composition (DXA) were taken and blood was collected prior to (PRE) and following the intervention period (POST). Blood samples were analyzed for monocyte cell-surface expression MC1R, MC3R, MC5R and C-reactive protein (CRP) and the plasma cytokines interleukin 6 (IL-6) and interleukin 10 (IL-10) using flow cytometry and ELISAs respectively.

ELIGIBILITY:
Inclusion Criteria:

* All Participants Must be Healthy
* The Strength Training Group Members Must Be Approved For Participation by a Licensed MD

Exclusion Criteria:

* Females may not be pregnant
* Unhealthy participants (those with existing conditions)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Melanocortin 1 Receptor Expression on Monocytes | Before and After 12 Week of Intervention Period
  Blood samples were analyzed for monocyte cell-surface expression of the melanocortin 1 receptor using flow cytometry. Pre samples were collected in Jan. 2010 and post samples were collected in May 2010 from all subjects.
Plasma CRP | Before and After the 12 Week Intervention Period
  Blood samples were analyzed for C-reactive protein using ELISA. Pre samples were collected in Jan. 2010 and post samples were collected in May 2010 from all subjects.
Body Composition (Fat Tissue Amount) | Before and After the 12 Week Intervention Period
  Body composition was assessed using DXA. Pre measures were completed in Jan. 2010 and post measures were completed in May 2010 for all subjects.
Plasma IL-6 | Before and After the 12 Week Intervention Period
  Blood samples were analyzed for IL-6 using ELISA. Pre samples were collected in Jan. 2010 and post samples were collected in May 2010 from all subjects.
Plasma IL-10 | Before and After the 12 Week Intervention Period
  Blood samples were analyzed for IL-10 using ELISA. Pre samples were collected in Jan. 2010 and post samples were collected in May 2010 from all subjects.
Melanocortin 3 Receptor Cell Surface Expression on Monocytes | Before and After the 12 Week Intervention Period
  Blood samples were analyzed for monocyte cell-surface expression of the melanocortin 3 receptor using flow cytometry. Pre samples were collected in Jan. 2010 and post samples were collected in May 2010 from all subjects.
Melanocortin 5 Receptor Cell Surface Expression on Monocytes | Before and After the 12 Week Intevention Period
  Blood samples were analyzed for monocyte cell-surface expression of the melanocortin 5 receptor using flow cytometry. Pre samples were collected in Jan. 2010 and post samples were collected in May 2010 from all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Laura K Stewart, PhD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- Louisiana State University, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Henagan TM, Forney L, Dietrich MA, Harrell BR, Stewart LK. Melanocortin receptor expression is associated with reduced CRP in response to resistance training. J Appl Physiol (1985). 2012 Aug;113(3):393-400. doi: 10.1152/japplphysiol.00107.2012. Epub 2012 Jun 7. PMID 22678961